CLINICAL TRIAL: NCT02052414
Title: Open Labeled, Non-randomized, Study of Efficacy and Safety of Gralise in Fibromyalgia Patients.
Brief Title: Study of Gralise to Treat Fibromyalgia Patients
Acronym: Gralise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Clinical Research, Winston-Salem, NC (Other)
Collaborators: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIR 2012-01
Record Dates: First submitted 2013-08-02; First posted 2014-02-03 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-09

CONDITIONS: Fibromyalgia
Keywords: side effects; safety; efficacy; Gralise; Fibromyalgia; gabapentin
MeSH Terms: conditions — Fibromyalgia | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gralise (Gabapentin ER) (Experimental): All patients will be treated with Gralise. Patients who are on pregabalin or gabapentin (lyrica or neurontin) will need to wash off the medication before starting Gralise.
  Patients who are ready to take Gralise will start with starter pack, and will gradually titrate the dose up to 1800mg per day. After that, patient will take 1800mg per day out of the bottle.
  Patient will be seen in clinic at 4weeks intervals for first 4 visits, and then there will be end of the study visit on week 15. On visit 4, week 12 of treatment, patients will be taught to taper off the study medication.
  Interventions: Drug: Gabapentin ER

INTERVENTIONS:
Drug: Gabapentin ER — Patient who are on gralise will report efficacy by rating his or her pain rating on a digital pain scale (11 points) from 0 to 10 on each scheduled clinical visits, which will be compared to their pain level at baseline.
  In addition, patients will also record the doses and any adverse effects that might arise during the trial in a diary provided by the study. All information will be recorded in a paper diary that will be followed by coordinator during each follow up visits.
  Other Names: Gralise

SUMMARY:
To determine Gralise in treating fibromyalgia pain:

* efficacy
* safety

DETAILED DESCRIPTION:
Subject must carry a diagnosis of fibromyalgia based on American College of Rheumatology (ACR) criteria for fibromyalgia

* Patient may be gaba-analogue (Pregabalin, trade name: lyrica, or Gabapentin, trade name: Neurontin) naïve, or had been on other gaba analogue before, and discontinued for lack of efficacy.
* Patient who had allergic reaction or serious adverse reactions will not be included in this study.
* Patient will start with starter pack of Gralise and will reach therapeutic dose of 1800 mg per day by end of 2 weeks.
* Drug is to be taken with meal, once a day in the evening; once patient has reached the therapeutic dose of 1800 mg, patient will come in for visit, at which point the PI will evaluate the patient and may increase or decrease the dosage, but patient may not increase or decrease the dose of medication at his /her discretion.
* During study, patient will have total of 5 visits, 4 of which will be for duration patient will be on Gralise, and the last visit will be for tapering off the medication.
* During study, patient is asked keep a paper diary on which patient will record the numeric pain scale from Fibromyalgia, time the medication was taken, dose of medication, and any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years and older.
* Subject carries Fibromyalgia diagnosis based on American College of Rheumatology criteria.
* Fibromyalgia patients who are gamma-aminobutyric acid (GABA)-analogue (gabapentin or pregabalin) naïve, or those who have been on gamma-aminobutyric acid (GABA)-analogue, but discontinued due to side effects or having difficulty maintaining dosing schedule due to multiple doses per day, or those who are currently on immediate release gamma-aminobutyric acid-analogue (GABA).
* Able to distinguish pain from fibromyalgia and pain from other sources. (subjects with other rheumatic disease or medical conditions that contributed to the symptoms of fibromyalgia will be excluded)
* Subject pain scores >4 on Numeric pain rating scale (NPRS)

Exclusion Criteria:

* Creatinine clearance of < 30mg/ml
* Pain from Traumatic injury or structural or regional rheumatic disease
* Unstable medical or psychiatric illness
* Lifetime history of psychosis, hypomania, or mania.
* Epilepsy, or dementia
* Substance abuse in the last 6 months
* Suicidal tendencies
* Pregnant or breastfeeding
* Not on contraception for those of childbearing age. (Barrier methods, oral contraception, hormone injections, or surgical sterilization)
* Subjects who are, in the opinion of the principle investigator, are treatment refractory
* Treatment with investigational drug within 30 days of screening.
* Concomitant medication exclusions consisted of medications or herbal agents with Central Nervous System (CNS) effects with exception of episodic use of sedating antihistamines
* Subject who are on more than one additional class of concomitant fibromyalgia medications i.e. non-selective serotonin reuptake inhibitor (SSRI) antidepressants, topicals, opioids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James North, MD, Principal Investigator — Center for Clinical Research
Locations (1):
- Center for Clinical Research, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No individual participants data will be shared with anyone who is not a member of the study staff, and all records containing individual data and their protected health information will remain confidential in accordance with the HIPAA rules.

REFERENCES:
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Hudson JI, Pope HG Jr. The relationship between fibromyalgia and major depressive disorder. Rheum Dis Clin North Am. 1996 May;22(2):285-303. doi: 10.1016/s0889-857x(05)70273-8. PMID 8860800
- [Background] Wolfe F, Ross K, Anderson J, Russell IJ, Hebert L. The prevalence and characteristics of fibromyalgia in the general population. Arthritis Rheum. 1995 Jan;38(1):19-28. doi: 10.1002/art.1780380104. PMID 7818567
- [Background] Arnold LM, Keck PE Jr, Welge JA. Antidepressant treatment of fibromyalgia. A meta-analysis and review. Psychosomatics. 2000 Mar-Apr;41(2):104-13. doi: 10.1176/appi.psy.41.2.104. PMID 10749947
- [Background] Arnold LM, Rosen A, Pritchett YL, D'Souza DN, Goldstein DJ, Iyengar S, Wernicke JF. A randomized, double-blind, placebo-controlled trial of duloxetine in the treatment of women with fibromyalgia with or without major depressive disorder. Pain. 2005 Dec 15;119(1-3):5-15. doi: 10.1016/j.pain.2005.06.031. Epub 2005 Nov 17. PMID 16298061
- [Background] Pillemer SR, Bradley LA, Crofford LJ, Moldofsky H, Chrousos GP. The neuroscience and endocrinology of fibromyalgia. Arthritis Rheum. 1997 Nov;40(11):1928-39. doi: 10.1002/art.1780401103. No abstract available. PMID 9365080
- [Background] Lautenbacher S, Rollman GB. Possible deficiencies of pain modulation in fibromyalgia. Clin J Pain. 1997 Sep;13(3):189-96. doi: 10.1097/00002508-199709000-00003. PMID 9303250
- [Background] Bennett RM. Emerging concepts in the neurobiology of chronic pain: evidence of abnormal sensory processing in fibromyalgia. Mayo Clin Proc. 1999 Apr;74(4):385-98. doi: 10.4065/74.4.385. PMID 10221469
- [Background] Staud R. Evidence of involvement of central neural mechanisms in generating fibromyalgia pain. Curr Rheumatol Rep. 2002 Aug;4(4):299-305. doi: 10.1007/s11926-002-0038-5. PMID 12126581
- [Background] Baranauskas G, Nistri A. Sensitization of pain pathways in the spinal cord: cellular mechanisms. Prog Neurobiol. 1998 Feb;54(3):349-65. doi: 10.1016/s0301-0082(97)00067-1. PMID 9481803
- [Background] Arnold LM, Goldenberg DL, Stanford SB, Lalonde JK, Sandhu HS, Keck PE Jr, Welge JA, Bishop F, Stanford KE, Hess EV, Hudson JI. Gabapentin in the treatment of fibromyalgia: a randomized, double-blind, placebo-controlled, multicenter trial. Arthritis Rheum. 2007 Apr;56(4):1336-44. doi: 10.1002/art.22457. PMID 17393438
- [Background] Gidal BE, DeCerce J, Bockbrader HN, Gonzalez J, Kruger S, Pitterle ME, Rutecki P, Ramsay RE. Gabapentin bioavailability: effect of dose and frequency of administration in adult patients with epilepsy. Epilepsy Res. 1998 Jul;31(2):91-9. doi: 10.1016/s0920-1211(98)00020-5. PMID 9714500
- See also: Drug manufacturer's website — http://depomed.com/
- See also: website for center for clinical research — http://www.centerforclinicalresearch.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Gralise (Gabapentin ER): An Open label trial with Gralise. All subjects on gabapentinoids will require wash before starting trial.
  All Subjects will follow the instructions on the Gralise starter pack with eventual goal of 1800 mg/day.
  Subjects will be have follow up visits every 4 weeks, and at the end of 12 weeks, subjects will begin to wash off of Gralise. Visit 5 will be end of the study/ treatment visit.
  Subject will rate pain ratings as primary outcome measure, and fibromyalgia impact questionnaires, medical study's outcome sleep scores, and patients global impression of change (PGIC) as secondary outcome measures. Subjects are assessed at each follow up visits for adverse events, and concomitant medication changes if any.
Period: Overall Study
Arm/Group | Gralise (Gabapentin ER)
Started | 34
Completed | 17
Not Completed | 17
Not completed — Adverse Event | 12
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Gralise (Gabapentin ER): This is an open label trial to evaluate the efficacy of Gralise against fibromyalgia pain. If subject is taking gabapentinoids at the time of enrollment, subjects will be required to wash off the medication; otherwise they can start the starter pack for Gralise, and will eventually up titrated to treatment dose of 1800mg with evening meals per day.
  Subjects will be followed every 4 weeks for total of 12 weeks. At the end of 12 weeks, subjects will be wash off the Gralise over 2 weeks, and will have a final end of treatment visit at week 15.
  Subjects will be asked to rate their pain on numeric pain rating system (NPRS) as primary outcome measure. Subjects will be asked to assess Fibromyalgia Impact Questionnaire (FIQ), Medical Outcome Study (MOS) Sleep questionnaire, and Patient Global Impression of Change (PGIC) as secondary outcome measures.
  At each follow up visits, occurrence of adverse events, and changes to concomitant medications were evaluated and recorded.
Arm/Group | Gralise (Gabapentin ER)
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.25 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 34
Age of Fibromyalgia Diagnosis [Mean (Full Range); unit: years] | 6.96 [1 to 7]
Number of active medications [Mean (Full Range); unit: medications] | 1.3 [1 to 2]
Number of past medications [Mean (Full Range); unit: medications] | 1.6 [0 to 7]
Number of co-morbid conditions [Mean (Full Range); unit: co-morbid conditions present] | 5.3 [2 to 14]
Gabapentinoid (Gabapentin/ pregabalin) Naive [Number; unit: participants] — Of all the subjects participated in this trial, 8 subjects were Gabapentinoid naïve.
  participants
    Gabapentinoid Naive | 8
    Non-Gabapentinoid naive | 26

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating System (NPRS)
Description: Fibromyalgia pain experienced by study subjects will be captured using NPRS at baseline visit, at each follow visits that are scheduled to occur every 4 weeks over 12 weeks of treatment period, and at the end of treatment visit that will occur 3 weeks after treatment period (12 weeks treatment period + 3 weeks = 15 weeks). Any difference in NPRS scores between baseline and any subsequent visits will indicate the magnitude of pain relief as reflected in digital scale of 0-10 (0=no pain, 10=worst pain imaginable).
Time Frame: 15 weeks
Population: All subjects had diagnosis of fibromyalgia and met the inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gralise (Gabapentin ER)
Number analyzed (Participants) | 31
units on a scale
  NPRS Baseline (Visit 1) | 7.29 (1.51)
  NPRS on Week 4 (Visit 2) | 4.72 (2.44)
  NPRS on week 8 (Visit 3) | 3.95 (2.18)
  NPRS on Week 12 (Visit 4) | 3.83 (2.05)
  NPRS on week 15 (Visit 5) | 6.94 (2.08)

2. Secondary Outcome: Medical Outcome Study (MOS) Sleep Questionnaires
Description: Medical Outcomes Study (MOS) sleep questionnaires to assess how Fibromyalgia impacts patients' sleep in various areas.
  Specifically, Data reported below measured number of hours subjects spent per night sleeping. MOS sleep questionnaires were assessed at each follow up visits. (visits 1, 2, 3, 4, and 5).
Time Frame: 15 weeks
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Gralise (Gabapentin ER)
Number analyzed (Participants) | 31
Hours
  Sleep Quantity Baseline | 5.86 (1.65)
  Sleep Quantity week 4 | 7.17 (1.62)
  Sleep quantity week 8 | 6.81 (1.81)
  Sleep quantity week 12 | 7.04 (0.72)
  Sleep quantity week 15 | 6.23 (1.71)

3. Secondary Outcome: Self Reported Side Effects.
Description: Side / adverse effects were assessed at each follow up visits and resulted are as follows.
Time Frame: 15 Weeks
Population: Subject who experienced pain, acute delirium, symptoms related to adhesions due to prior surgical procedures, extremity swelling, and possible drug interactions discontinued medications. Other reported side effects dissipated after subjects reached therapeutic dose of 1800mg of study medication taken at bedtime.
Measure: Number; unit: participants
Groups:
- Gralise (Gabapentin ER): All subjects were assessed for occurrence of adverse events at follow up visits. All reported adverse events were tabulated, and presented in this study.
Arm/Group | Gralise (Gabapentin ER)
Number analyzed (Participants) | 31
participants
  Extremity Swelling | 2
  Weight Gain | 2
  Drowsy | 8
  Dizzy | 3
  Irritability | 3
  Dry Eyes | 2
  Pain | 1
  Mood Changes | 2
  Difficulty Concentrating | 2
  Dry Mouth | 1
  Suspected Drug interaction | 1
  Acute Delerium | 1
  Adhesion | 1
  None | 12

4. Secondary Outcome: Fibromyalgia Impact Questionnaire (FIQ)
Description: The Fibromyalgia Impact Questionnaire (FIQ) is an instrument designed to quantitate the overall impact of fibromyalgia over many dimensions (e.g. function, pain level, fatigue, sleep disturbance, psychological distress etc.). It is scored from 0 to 100 with the latter number being the worst case. The average score for patients seen in tertiary care settings is about 50. The FIQ is widely used to assess change in fibromyalgia status.
Time Frame: 15 weeks.
Population: FM patients who took study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gralise (Gabapentin ER)
Number analyzed (Participants) | 31
units on a scale
  FIQ Baseline | 71.04 (12.84)
  FIQ Week 4 | 41.82 (19.57)
  FIQ Week 8 | 40.79 (20.41)
  FIQ Week 12 | 39.27 (21.37)
  FIQ Week 15 | 61.86 (18.67)

5. Other Pre Specified Outcome: Patient Global Impression of Change (PGIC)
Description: Patient Global impression of Change (PGIC) is an outcome commonly used measure of the efficacy of treatments. PGIC is a 7 point scale that requires the subjects to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: 15 Weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gralise (Gabapentin ER)
Number analyzed (Participants) | 31
units on a scale
  PGIC After 4 weeks | 4.96 (1.61)
  PGIC After 8 weeks | 5.40 (1.31)
  PGIC After 12 weeks | 5.37 (1.54)
  PGIC After 15 weeks | 4.44 (1.97)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected at baseline (visit 1), week 4 (visit 2), week 8 (visit 3), week 12 (visit 4), and week 15 (visit 5). If subject required unscheduled visit, AE were collected as part of the visit procedure.
Arm/Group | Gralise (Gabapentin ER)
Serious Adverse Events (participants affected / at risk) | 2/31
Other Adverse Events (participants affected / at risk) | 10/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gralise (Gabapentin ER) (N=31)
Small bowel adhesion (Gastrointestinal disorders) | 1 (1) — Subject had a laparoscopic bariatric surgery few years ago, and as a consequence subject suffered a bowel adhesion and subsequent small bowel obstruction. Subject underwent lysis of adhesion, and recovered without sequelae.
Acute Delirium (Nervous system disorders) | 1 (1) — Subject exhibited early signs and symptoms of alzheimers symptoms. Subject was seen at ED on Friday, and admitted to neurology care for observation and work up over the weekend. \
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gralise (Gabapentin ER) (N=31)
Extremity swelling (Metabolism and nutrition disorders) | 2 (2) — bilateral upper extremity swelling.
Weight Gain (Metabolism and nutrition disorders) | 2 (2) — Subjects gained weight after starting on study medication
Drowsiness (Nervous system disorders) | 8 (8) — Drowsy
Dizzines (Ear and labyrinth disorders) | 3 (3) — Dizzy
irritability (Psychiatric disorders) | 3 (3)
dry eyes (Eye disorders) | 2 (2)
pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Mood changes (Psychiatric disorders) | 2 (2)
Difficulty Concentrating (Nervous system disorders) | 2 (2)
drymouth (Gastrointestinal disorders) | 1 (1)
drug interaction (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
small sample size, geographical bias, relatively short duration of treatment, open label, single arm study without a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No